CLINICAL TRIAL: NCT03984279
Title: Comparison of the Study Was to Compare Sequential Fluoroscopy Guidance With Spiral Guidance in Terms of Safety (Number of Major Complications), Effectiveness (Number of Targets Reached), Speed (Procedural Time) and Radiation (DLP) in Interventional Chest-abdomen-pelvic Procedures.
Brief Title: Comparison of Sequential Fluoroscopy Guidance With Spiral Guidance in Terms of Safety, Effectiveness, Speed and Radiation in Interventional Chest-abdomen-pelvic Procedures
Acronym: APIR-TDM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2018/362
Record Dates: First submitted 2019-05-27; First posted 2019-06-12 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-05

CONDITIONS: Body Interventional procédures With CT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sequentiel group (SEQ)
  Interventions: Other: Patients with indication of interventional percutaneous diagnostic or therapeutic chest-abdomen-pelvic procedure under CT control
- Siral group (SPI)
  Interventions: Other: Patients with indication of interventional percutaneous diagnostic or therapeutic chest-abdomen-pelvic procedure under CT control

INTERVENTIONS:
Other: Patients with indication of interventional percutaneous diagnostic or therapeutic chest-abdomen-pelvic procedure under CT control — Not applicable, all patients with indication of interventional percutaneous diagnostic or therapeutic chest-abdomen-pelvic procedure under CT control on a period of 1 year will be taken into account

SUMMARY:
The purpose of the study was to compare sequential fluoroscopy guidance with spiral guidance in terms of safety (number of major complications), effectiveness (number of targets reached), speed (procedural time) and radiation (DLP) in interventional chest-abdomen-pelvic procedures.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (> 18 years),
* indication of interventional percutaneous diagnostic or therapeutic chest-abdomen-pelvic procedure under CT control

Exclusion Criteria:

* MRI contra indication
* persons referred to in Articles L1121-5 to L1121-8 of the French Public Health Code

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with indication of interventional percutaneous diagnostic or therapeutic chest-abdomen-pelvic procedure under CT control
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
number of major complications | All patients with indication of interventional percutaneous diagnostic or therapeutic chest-abdomen-pelvic procedure under CT control performed on a period of 1 year will be taken into account
  Comparison between the 2 groups
number of targets reached | All patients with indication of interventional percutaneous diagnostic or therapeutic chest-abdomen-pelvic procedure under CT control performed on a period of 1 year will be taken into account
  Comparison between the 2 groups
Dose Length Product (DLP) | All patients with indication of interventional percutaneous diagnostic or therapeutic chest-abdomen-pelvic procedure under CT control performed on a period of 1 year will be taken into account
  Comparison between the 2 groups

SECONDARY OUTCOMES:
number of controls required to place the needle | All patients with indication of interventional percutaneous diagnostic or therapeutic chest-abdomen-pelvic procedure under CT control performed on a period of 1 year will be taken into account
  Comparison between the 2 groups

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Besançon, France